CLINICAL TRIAL: NCT02380378
Title: Registry of Philadelphia-Negative Myeloproliferative Neoplasms
Acronym: MPN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Hospital Santa Marcelina (Other); Instituto Nacional de Cancer, Brazil (Other Government); Federal University of Minas Gerais (Other); Irmandade da Santa Casa de Misericordia de Sao Paulo (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Fabio Pires de Souza Santos, Fabio Pires de Souza Santos, Hospital Israelita Albert Einstein
Other Study IDs: RMPN2015
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Myeloproliferative Neoplasms: Patients diagnosed with Myeloproliferative Neoplasms based on WHO 2008 criteria.

SUMMARY:
This study was developed to document current diagnosis and treatment patterns, clinical outcomes, and health care resource use associated with Philadelphia-Negative Myeloproliferative Neoplasms, in the different risk classifications for each disease.

DETAILED DESCRIPTION:
Philadelphia-negative (Ph-negative) Myeloproliferative Neoplasms (MPN) include polycythemia vera (PV), essential thrombocythemia (TE), and primary myelofibrosis (MF). Ph-negative MPN are chronic myeloid neoplasms that appear after a malignant transformation of a hematopoietic stem cell. There are many clinical manifestations of these diseases, which include polyglobulia, thrombocytosis, leukocytosis, cytopenias, extramedullary hematopoiesis (e.g.: splenomegaly), increased thrombotic risk and the risk of transformation to acute myeloid leukemia (AML). Life expectancy varies from 5-6 years for patients with MF to more than 15 years for patients with PV and ET.

There are few therapeutic options for patients with Ph-negative MPN. In general, the treatment of these diseases is symptomatic and targeted to the relief of symptoms and control of hematological setting using oral chemotherapy agents such as hydroxyurea. Patients with MF receive palliative treatment, targeted to the relief of splenomegaly and cytopenias. Currently, there are no approved drugs for the treatment of MF.

In Latin America, there are no epidemiological studies with a great number of Ph-negative MPN patients describing the natural history of the disease, patient progress, clinical characteristics, standards of care and disease burden. The development of an up-to-date data registry of Brazilian patients with Ph-negative MPN allows the comprehension of the epidemiology of this disease, with determination of survival, thrombosis incidence, transformation to AML, use of disease treatment-related resources, as well as the impact of different therapeutic strategies in these parameters. Therefore, the objective of this study is to establish a registry of patients with Ph-negative MPN in order to document the disease diagnosis and current standards of care, clinical endpoints, and the use of treatment-related resources, according to risk classification in each MPN.

Data will be retrospectively and prospectively collected through an electronic form available at an Internet safe website. Each center participating in the study will have a principal investigator who will be in charge of the accuracy and quality of the data collected. Each principal investigator and staff will receive a login and a password to access the database and enroll patients in the registry. An employee from each site will be in charge of collecting the data and inserting them in the electronic registry. Patients shall be contacted in order to sign an informed consent form. Patient data will be updated every six months. There is no limit for the number of patients to be enrolled in the registry, either retrospectively or prospectively. The duration of this study is five years. Data collection will continue until all sites decide to interrupt the enrollment of new patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of (according to WHO 2008 criteria) Polycythemia Vera, Essential Thrombocythemia, Primary Myelofibrosis or Post-Polycythemia Vera/Post-Essential Thrombocythemia Myelofibrosis, Unclassifiable Myeloproliferative Neoplasm, Chronic Neutrophilic Leukemia, Chronic Eosinophilic Leukemia, Systemic Mastocytosis
* diagnosis made since 2000
* patients who are being followed-up or not
* signed informed consent form (for alive patients included in the prospective step of the study).

Exclusion Criteria:

* diagnosis of Chronic Myelogenous Leukemia
* refusal to sign the informed consent form (for patients who are alive and will de included in the prospective step of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are followed in hematological centers with confirmed diagnosis of Myeloproliferative Neoplasms since 2000.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2022-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Registry of Philadelphia-Negative Myeloproliferative Neoplasms | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Fabio P Santos, Principal Investigator — Instituto Israelita de Ensino e Pesquisa Albert Einstein´s (IIEP)
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil